CLINICAL TRIAL: NCT02932020
Title: Pilot Study Investigating the Utility of Epidural AlloGen-LI Injection for Treatment of Spinal Stenosis Symptoms
Brief Title: AlloGen-LI Treatment of Spinal Stenosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: VIVEX Biologics, Inc. (Industry)
Responsible Party: Principal Investigator, Wende Gibbs, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HS-15-00576
Record Dates: First submitted 2016-10-04; First posted 2016-10-13 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Low Back Pain
Keywords: disc herniation; spinal stenosis
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement; Spinal Stenosis | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Randomized 10 subjects
  Visit 1:
  1st contrast enhanced Magnetic Resonance Imaging (MRI) scan of the lumbar spine interlaminar epidural injection of (a) 2mL 0.5% marcaine and one 2-ml dose of AlloGen-LI
  Visit: 6 weeks (+7days): 2nd contrast enhanced Magnetic Resonance Imaging (MRI) scan of the lumbar spine
  Interventions: Drug: AlloGen-LI; Device: MRI; Drug: 0.5% marcaine
- Group B (Other): Randomized 10 subjects
  Visit 1:
  1st contrast enhanced Magnetic Resonance Imaging (MRI) scan of the lumbar spine interlaminar epidural injection 2mL 0.5% marcaine and 1mL and 1mL steroid (depomedrol 80mg/ml).
  Visit 6 weeks (+7days): 2nd contrast enhanced Magnetic Resonance Imaging (MRI) scan of the lumbar spine
  Interventions: Drug: depomedrol; Device: MRI; Drug: 0.5% marcaine

INTERVENTIONS:
Drug: AlloGen-LI — interlaminar epidural injection of 2mL 0.5% marcaine and one 2-ml dose of AlloGen-LI
  Other Names: Interlaminar Epidural Injection-AlloGen-LI
  Arms: Group A
Drug: depomedrol — interlaminar epidural injection of 2mL 0.5% marcaine and 1mL steroid (depomedrol 80mg/ml)
  Other Names: Interlaminar Epidural Injection-Standard
  Arms: Group B
Device: MRI — contrast enhanced MRI of the lumbar spine performed at Visit 1 and Visit 6 weeks (+7 days)
Drug: 0.5% marcaine — epidural injection of 2mL 0.5% marcaine

SUMMARY:
In this pilot study, investigators will test the efficacy of AlloGen-LI, an allograft derived from amniotic fluid, injected into the epidural space at the level of spinal stenosis as an anti-inflammatory treatment to relieve back and leg pain symptoms in patients with spinal stenosis and/or disc herniation. The patients will be followed for 12 weeks. The effect of this treatment will be examined by patient reported changes in pain and disability utilizing validated outcome measures, and MRI imaging evaluating changes in contrast enhancement and T2 signal related to that reflect inflammation and degeneration.

DETAILED DESCRIPTION:
AlloGen-LI contains multiple factors that may serve to ameliorate the detrimental effects of osteorarthritis and degenerative disc disease. Anti-inflammatory components include inhibitors of matrix metalloproteins and pro-inflammatory cytokines, growth factors and interleukins. The product has low immunogenicity and is hypo-osmotic.2 Placental tissues, including amniotic fluid, amniotic membrane and chorion are regulated as human cell and tissue products (HCTP) by the FDA. This regulation allows clinicians to use the allograft materials for human injection. AlloGen-LI is derived from placental tissues obtained from carefully screened healthy mothers at the time of scheduled cesarean section. The mothers have agreed to donate the tissues, which would otherwise be discarded. The experimental treatment would entail an injection of one dose of AlloGen-LI and marcaine into the epidural space under CT guidance, in an identical manner to traditional epidural steroid /marcaine injections.

ELIGIBILITY:
Inclusion Criteria:

1. Low back pain of > 4-5 weeks but < 6-7 months
2. Evidence of at least mild lumbar stenosis /disc herniation on MRI
3. Failure of conservative therapy to include physical therapy and pharmacotherapy
4. Patient is at least 18 years of age
5. Patient is willing to be blinded to treatment until after the 12 week post injection visit
6. Patient is willing and able to review and sign the study informed consent form

Exclusion Criteria:

1. No evidence of lumbar stenosis or disc herniation on MRI 2. Patient has had prior lumbar surgery at any level 3. Patient has received epidural steroid injection in the past 6 months 4. Patient currently receives systemic steroids for another medical condition 5. Patient is pregnant 6. Patient has systemic infection at the proposed injection site 7. Patient has a systemic malignancy 8. Current therapy with any immunosuppressive medication 9. History of solid organ or hematologic transplantation 10 History of autoimmune disorder 11. Patient has known allergy to lidocaine, marcaine or steroid 12. Devices and conditions that are contraindications for MRI examination (routinely screened before all MRI examinations).

13. Patient is on anticoagulant medications (other than ASA). 14. Patient has eGFR of <40 15. Patient has known chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | 6-12 weeks
  Cohen's d25 will be calculated at each permutation iteration. The empirical distribution of Cohen's d will then be calculated with a 95% confidence interval (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Wende Gibbs, MD, Principal Investigator — University of Southern California
Locations (1):
- Keck School of Medicine of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided